CLINICAL TRIAL: NCT00349024
Title: Efficacy of Gelclair™ in Reducing the Pain of Oral Mucositis in Children and Young People With Cancer (SC 2005 07)
Brief Title: Polyvinylpyrrolidone-Sodium Hyaluronate Gel in Reducing Pain From Oral Mucositis in Young Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000481526; CCLG-SC-2005-07; EU-20621
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors; Chordoma; Kidney Cancer; Leukemia; Lymphoma; Mucositis; Neuroblastoma; Pain; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; pain; childhood acute lymphoblastic leukemia; childhood Hodgkin lymphoma; chondrosarcoma; osteosarcoma; childhood soft tissue sarcoma; Wilms tumor and other childhood kidney tumors; neuroblastoma; childhood acute myeloid leukemia/other myeloid malignancies; childhood large cell lymphoma; childhood lymphoblastic lymphoma; childhood small noncleaved cell lymphoma; childhood rhabdomyosarcoma; childhood brain stem glioma; childhood central nervous system germ cell tumor; childhood cerebellar astrocytoma; childhood cerebral astrocytoma/malignant glioma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood ependymoma; childhood medulloblastoma; childhood meningioma; childhood oligodendroglioma; childhood atypical teratoid/rhabdoid tumor; childhood spinal cord neoplasm; childhood supratentorial primitive neuroectodermal tumor; childhood visual pathway and hypothalamic glioma; chordoma; mucositis; Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Central Nervous System Neoplasms; Chordoma; Kidney Neoplasms; Leukemia; Lymphoma; Mucositis; Neuroblastoma; Pain; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Chondrosarcoma; Osteosarcoma; Wilms Tumor; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Medulloblastoma; Meningioma; Oligodendroglioma; Rhabdoid Tumor; Spinal Cord Neoplasms; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Gelclair

INTERVENTIONS:
Drug: polyvinylpyrrolidone-sodium hyaluronate gel

SUMMARY:
RATIONALE: Polyvinylpyrrolidone-sodium hyaluronate gel may lessen the pain of oral mucositis, or mouth sores, in patients undergoing treatment for cancer.

PURPOSE: This clinical trial is studying how well polyvinylpyrrolidone-sodium hyaluronate gel works in reducing pain from oral mucositis in young patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the feasibility and acceptability of polyvinylpyrrolidone-sodium hyaluronate gel in pediatric patients experiencing oral pain from mucositis after cancer therapy.

OUTLINE: This is a prospective, uncontrolled, open-label, pilot, multicenter study.

Beginning before hospital discharge or day 3 after chemotherapy, patients use oral polyvinylpyrrolidone-sodium hyaluronate gel mouth rinse for at least 1 minute, 3 times per day or as needed. Treatment continues for 48 hours. Patients with persistent oral pain may continue treatment with polyvinylpyrrolidone-sodium hyaluronate gel beyond 48 hours.

Oral pain and acceptability (i.e., taste) of polyvinylpyrrolidone-sodium hyaluronate gel are assessed periodically using self-reported rating scales.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer, including, but not limited to, the following:

  * Acute lymphoblastic leukemia
  * Acute myeloid leukemia
  * Brain tumor
  * Hodgkin's lymphoma
  * Non-Hodgkin's lymphoma
  * Sarcoma
  * Wilms' tumor
  * Neuroblastoma
* Meets 1 of the following criteria:

  * Admitted to an in-patient unit after undergoing chemotherapy that is anticipated to cause oral mucositis
  * Admitted to an in-patient unit after undergoing myeloablative therapy followed by peripheral blood stem cell or bone marrow transplantation
* Is experiencing oral pain due to mucositis

PATIENT CHARACTERISTICS:

* No known hypersensitivity to polyvinylpyrrolidone-sodium hyaluronate gel

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent analgesics allowed

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Timing and intensity of oral pain
Duration of action of polyvinylpyrrolidone-sodium hyaluronate gel
Acceptability, effectiveness, and adherence to regimens including polyvinylpyrrolidone-sodium hyaluronate gel
Symptoms, other than pain, considered important to the pediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gibson, MD — Great Ormond Street Hospital for Children NHS Foundation Trust; Tim O.B. Eden, MB, BS, FRCPE, FRCP, FRCPCH, F — The Christie NHS Foundation Trust
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales